CLINICAL TRIAL: NCT04778423
Title: AVATAR Therapy to Reduce the Power of the Eating Disorder Voice in Eating Disorders: Collaborative Development and Feasibility Testing
Brief Title: Feasibility and Acceptability of AVATAR Therapy in Eating Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 292346
Record Dates: First submitted 2021-02-19; First posted 2021-03-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-02

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avatar Therapy (Experimental): AVATAR therapy for eating disorders
  Interventions: Other: Avatar Therapy

INTERVENTIONS:
Other: Avatar Therapy — In the first session (assessment), participants will create a computerised representation of the eating disorder voice (avatar) on a computer. They will be able to manipulate the facial and voice characteristics of the avatar and will be asked to provide examples of the critical eating disorder comments most often spoken by the avatar. In the following sessions (6-8 therapy sessions), participants will interact with the avatar displayed on the computer screen for 5-10 minutes.The main goal during the interaction with the avatar is for participants to stand up to the critical comments made by the avatar and build a sense of power, control and self-awareness in the context of the eating disorder voice. The sessions will be conducted remotely, using a personal laptop or computer. This will provide patients with the opportunity to practise answering back to the eating disorder voice during a meal, a time at which the eating disorder voice is loudest.

SUMMARY:
This project will answer the overarching research question "What is the feasibility of developing and implementing AVATAR therapy to reduce the power of the eating disorder voice in patients with eating disorders?". AVATAR therapy for eating disorders has been developed based on AVATAR therapy for psychosis. The feasibility of using AVATAR therapy in eating disorders will be tested using non-concurrent multiple baselines single case experimental design. The first stage (A1) will involve participants being randomly allocated to either a two, three or four week-baseline. The second will be the intervention phase (B) where participants will receive the AVATAR treatment which will last approximately 6 weeks. The third stage (A2) will be a 4-week follow-up period after the intervention phase, where participants will also complete a qualitative interview.

DETAILED DESCRIPTION:
This project will answer the overarching research question "What is the feasibility of developing and implementing AVATAR therapy to reduce the power of the eating disorder voice in patients with eating disorders?". The aims are: 1) To use a collaborative approach that involves patients, carers and clinicians to adapt the AVATAR therapy in psychosis for patients with eating disorders. 2) To assess the feasibility of using this therapy in eating disorders.

Aim 1. To use a collaborative approach that involves patients, carers and clinicians to adapt the AVATAR therapy in psychosis for patients with eating disorders

Methods: Two collaborative workshops will be organised with a total of 16 people with lived experience of the illness (patients or carers) and 16 clinicians (approximately eight people/workshop), to review the contents of AVATAR therapy for eating disorders developed based on AVATAR therapy for psychosis. We will describe the structure and content of the therapy manual and will encourage the members of the group to provide feedback. The workshop will be video recorded. We will revise the therapy manual based on an iterative process of feedback and review. Outcome: the outcome will consist of a revised version of the AVATAR therapy manual.

Aim 2. To assess the feasibility of using AVATAR therapy in eating disorders

General procedure

Participants will be recruited through online advertisements and flyers placed at South London and Maudsley Hospital NHS Trust. They will be able to contact the researchers involved in the study by email. The researchers will then send the study information sheet by email and will assess eligibility to take part, should the participants wish to take part. Once eligibility is confirmed, participants will received a link to Qualtrics. Survey settings will eliminate the possibility of missing or repeated data. Participants will freely access the survey via a web link on the Internet. The online survey will include completion of the baseline questionnaires (described below). At the end of the intervention, and four-week follow-up, participants will receive two more links to Qualtrics, to complete the end-of-intervention and follow-up questionnaires, respectively. Following completion of the baseline questionnaires, participants will be invited to take part in the AVATAR therapy (described below), which will be delivered by one of the clinical researchers in the team. AVATAR therapy will be delivered remotely using a secure encrypted video-call system which will enable the delivery of the therapy in accordance with the clinical manual.

Design The project will use a non-concurrent multiple baselines single case experimental design (SCED) divided into three stages (A1BA2). The first stage (A1) will involve participants being randomly allocated to either a two, three or four week-baseline. The second will be the intervention phase (B) where participants will receive the AVATAR treatment which will last approximately 6 weeks. The third stage (A2) will be a 4-week follow-up period after the intervention phase, where participants will also complete a qualitative interview. Participants will be randomly allocated to variable baselines using a random number generator.

Sample size justification

We propose collecting data from 50 individuals. This is supported by scholars who suggest numbers ranging from 24 to 50 for feasibility studies.

AVATAR therapy for eating disorders

The therapy will be delivered by the members of the research team. In the first session (assessment), following a clinical assessment of the role of the eating disorder voice, participants will create a computerised representation of the eating disorder voice (avatar) on a computer. They will be able to manipulate the facial and voice characteristics of the avatar and will be asked to provide examples of the critical eating disorder comments most often spoken by the avatar. In the following sessions (6-8 therapy sessions), participants will interact with the avatar displayed on the computer screen for 5-10 minutes. The therapist will facilitate the dialogue by speaking the avatar's voice as well as their own (therapist) voice from a different room. The therapist will have a video link with the participant and therefore will be able to monitor the participants' responses to the avatar. The participant will be able to press a "stop" button should they want to stop the session. The main goal during the interaction with the avatar is for participants to stand up to the critical comments made by the avatar and build a sense of power, control and self-awareness in the context of the eating disorder voice. The sessions will be conducted remotely, using a personal laptop or computer. This will provide patients with the opportunity to practise answering back to the eating disorder voice during a meal, a time at which the eating disorder voice is loudest. The content of the sessions has been adapted from AVATAR for psychosis and is subject to further review as outlined in Research Aim 1.

Feasibility outcomes

(1) Recruitment of 80% or more of the targeted sample size in 18 months, (2) Adherence to protocol: 80% retention rate at 6-8 weeks (end of therapy), (3) Adherence to AVATAR therapy: 80% of patients completing at least 5 sessions (based on average attendance of 5 sessions in the psychosis trial), (4) Participants' satisfaction with the AVATAR therapy (80% of participants reporting a satisfaction rating of 7 or over, on a Likert scale ranging from 0 "not satisfied at all" to 10 "very satisfied"), (5) Estimation of effect size and standard deviation of change in power of the eating disorder voice and eating disorder symptoms. In addition to these parameters, we will record any issues related to the technical functioning or operation of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of anorexia nervosa or atypical anorexia nervosa (e.g. restored weight but presence of abnormal eating disorder cognitions and behaviors), bulimia nervosa or binge eating disorder
* availability of a laptop and internet connection for the assessments and sessions

Exclusion Criteria:

* diagnosis of psychosis, alcohol use disorder, substance use disorder
* insufficient level of English to engage in the therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of AVATAR therapy for eating disorder | 18 months
  Recruitment of 80% or more of the targeted sample size in 18 months and 80% retention to the study protocol at 6-8 weeks (end of therapy).

SECONDARY OUTCOMES:
Adherence | 18 months
  Adherence to AVATAR therapy: 80% of patients completing at least 5 sessions (based on average attendance of 5 sessions in the psychosis's trial)
Acceptability | 18 months
  Participants' satisfaction with the AVATAR therapy (80% of participants reporting a satisfaction rating over 7, on a Likert scale ranging from 0 "not satisfied at all" to 10 "very satisfied"
Eating disorder voice characteristics | 12 to 15 weeks depending on the baseline allocation
  Estimation of effect size and standard deviation of change in power of the eating disorder voice which will be measured by the auditory hallucination subscale of the psychotic symptom rating scale adapted for eating disorders, the beliefs about the voices questionnaires adapted for eating disorders and a brief weekly survey to assess the content and perceived power of the eating disorder voice.
Eating disorder symptoms | 12 to 15 weeks depending on the baseline allocation
  Eating disorder symptoms will be measured by the Eating disorder examination questionnaire (EDE-Q)
Anxiety and depression | 12 to 15 weeks depending on the baseline allocation
  Measured by the Depression, Anxiety and stress scales (DASS-21)
Self-criticism and self-compassion | 12 to 15 weeks depending on the baseline allocation
  Measured by self-criticism and self-compassion scale

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

REFERENCES:
- [Background] Noordenbos G, Aliakbari N, Campbell R. The relationship among critical inner voices, low self-esteem, and self-criticism in eating disorders. Eat Disord. 2014;22(4):337-51. doi: 10.1080/10640266.2014.898983. Epub 2014 Mar 28. PMID 24678635
- [Background] Pugh M, Waller G. The anorexic voice and severity of eating pathology in anorexia nervosa. Int J Eat Disord. 2016 Jun;49(6):622-5. doi: 10.1002/eat.22499. Epub 2016 Feb 15. PMID 26875724
- [Background] Falconer CJ, King JA, Brewin CR. Demonstrating mood repair with a situation-based measure of self-compassion and self-criticism. Psychol Psychother. 2015 Dec;88(4):351-65. doi: 10.1111/papt.12056. Epub 2015 Feb 5. PMID 25663161
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Craig TK, Rus-Calafell M, Ward T, Leff JP, Huckvale M, Howarth E, Emsley R, Garety PA. AVATAR therapy for auditory verbal hallucinations in people with psychosis: a single-blind, randomised controlled trial. Lancet Psychiatry. 2018 Jan;5(1):31-40. doi: 10.1016/S2215-0366(17)30427-3. Epub 2017 Nov 23. PMID 29175276
- [Derived] Thompson A, Calissano C, Treasure J, Ball H, Montague A, Ward T, Cardi V. A case series to test the acceptability, feasibility and preliminary efficacy of AVATAR therapy in anorexia nervosa. J Eat Disord. 2023 Oct 13;11(1):181. doi: 10.1186/s40337-023-00900-1. PMID 37833732